CLINICAL TRIAL: NCT07110584
Title: A Phase 1/2, Multi-Center, Open-Label Clinical Study Evaluating MDX2004 In Participants With Advanced Tumors
Brief Title: Dose Escalation and Dose Expansion Study of MDX2004 in Participants With Advanced Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ModeX Therapeutics, An OPKO Health Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MDX-2004-101
Record Dates: First submitted 2025-07-24; First posted 2025-08-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-11

CONDITIONS: Advanced Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose Escalation - Part A (Experimental): Participants with advanced tumors will receive MDX2004 as intravenous (IV) infusion.
  Interventions: Drug: MDX2004
- Indication Optimization - Part B (Experimental): Participants with select advanced tumors will receive MDX2004 as intravenous (IV) infusion.
  Interventions: Drug: MDX2004
- Dose Optimization - Part C (Experimental): Participants with select advanced tumors will receive one of two recommended doses of MDX2004 as intravenous (IV) infusion.
  Interventions: Drug: MDX2004
- Dose Expansion - Part D (Experimental): Participants with select advanced tumors will receive the recommended Phase 2 dose of MDX2004 as intravenous (IV) infusion.
  Interventions: Drug: MDX2004

INTERVENTIONS:
Drug: MDX2004 — MDX2004 intravenous infusion

SUMMARY:
This study is designed to characterize the safety, tolerability, and anti-tumor activity of MDX2004 in patients with advanced tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 years of age.
* Histologically or cytologically confirmed diagnosis of locally advanced or metastatic malignancy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* All participants should have at least 1 measurable site of disease according to RECIST v1.1. An irradiated lesion can be considered measurable only if progression has been demonstrated on the irradiated lesion.
* Adequate hematologic, hepatic and renal function.
* All contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Any clinically significant cardiac disease.
* Unresolved toxicities from previous anticancer therapy.
* Known untreated, active, or uncontrolled brain metastases.
* Previous Grade 3 or 4 immune-related toxicity that led to the discontinuation of treatment, within 6 months prior to the first dose of MDX2004.
* Active medical condition requiring chronic systemic steroid use (>10 mg/day prednisone or equivalent) or immunosuppressive therapy, within 6 months prior to the first dose of MDX2004.
* Known positivity with human immunodeficiency virus (HIV), known active hepatitis B or C, or uncontrolled chronic or ongoing infection requiring intravenous treatment.
* Prior solid organ or hematologic transplant
* Require supplemental oxygen for activities of daily living
* Participant is not suitable for participation, whatever the reason, as judged by the Investigator including medical or clinical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2031-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
All Study Parts: Adverse Events (AEs) | Baseline until 90 days after the participant has the last dose of MDX2004
  Incidence and severity of adverse events (AEs) and serious AEs (SAEs), including changes in clinical laboratory parameters, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.0 or American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading criteria, including changes in clinical laboratory parameters
Part A only - Maximum Tolerated Dose (MTD) or Recommended Phase 2 dose (RP2D) | 28 days
  Maximum Tolerated Dose or Recommended Phase 2 dose is determined following the evaluation of MDX2004 safety including the incidences of dose limiting toxicities (DLTs), MDX2004 anti-tumor activity, and MDX2004 pharmacokinetics/pharmacodynamics.
Part B, C, and D: Objective response rate of MDX2004 | From date of enrollment until the end of treatment, up to approximately 6 months
  Objective response rate is defined as the proportion of patients who achieve a complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
All Study Parts: Measure of terminal half-life (t1/2) of MDX2004 | 6 months
  Characterize pharmacokinetic (PK) parameter t1/2 after intravenous infusion of MDX2004.
All Study Parts: Measure of area under the serum concentration-time curve (AUC) of MDX2004 | 6 months
  Characterize pharmacokinetic (PK) parameter AUC after intravenous infusion of MDX2004
All Study Parts: Measure of time to maximum concentration (Tmax) of MDX2004 | 6 months
  Characterize pharmacokinetic (PK) parameter Tmax after intravenous infusion of MDX2004
All Study Parts: Measure of maximum serum concentration (Cmax) of MDX2004 | 6 months
  Characterize pharmacokinetic (PK) parameter Cmax after intravenous infusion of MDX2004
All Study Parts: Measure of volume of distribution (Vd) of MDX2004 | 6 months
  Characterize pharmacokinetic (PK) parameter Vd after intravenous infusion of MDX2004.
All Study Parts: Measure of system clearance of MDX2004 | 6 months
  Characterize pharmacokinetic (PK) parameter of system clearance after intravenous infusion of MDX2004.
All Study Parts: Evaluation of MDX2004 immunogenicity | 6 months
  The presence and persistence of anti-MDX2004 antibodies.
All Study Parts: Pharmacodynamic characterization of MDX2004 | 6 months
  Changes in T cell phenotypes with MDX2004 administration within the tumor microenvironment (TME) and in blood
All Study Parts: Duration of Response (DoR) | From date of enrollment until the end of treatment, up to approximately 6 months
  Time from first Complete Response (CR) / Partial Response (PR) to the date of progressive disease (PD) or death, whichever occurs first.
All Study Parts: Time to Response | From date of enrollment until the end of treatment, up to approximately 6 months
  The time from first dose to first documentation of response (CR or PR).
All Study Parts: Disease Control Rate (DCR) | From date of enrollment until the end of treatment, up to approximately 6 months
  The proportion of evaluable participants with stable disease (SD) or a best overall response of CR or PR.
All Study Parts: Progression Free Survival (PFS) | From date of enrollment until the end of treatment, up to approximately 6 months
  The time from the first dose of MDX2004 until the date of disease progression (PD) or death (any cause), whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (2):
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
- Israel (3):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv